CLINICAL TRIAL: NCT03375580
Title: Therapeutic Effects of Compound Zhenzhu Tiaozhi Capsules in Nonalcoholic Fatty Liver disease-a Randomized Controlled Study
Brief Title: Therapeutic Effects of Compound Zhenzhu Tiaozhi Capsules in NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Principal Investigator, He Xingxiang, Director of the Hospital, The First Affiliated Hospital of Guangdong Pharmaceutical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1201-8245
Record Dates: First submitted 2017-11-26; First posted 2017-12-18 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Metformin; Simvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TLC group (Placebo Comparator): transform life custom (TLC) group
  Interventions: Dietary Supplement: TLC
- TLC + metformin group (Active Comparator): transform life custom (TLC) combined with 0.5g metformin, PO tid
  Interventions: Dietary Supplement: TLC; Drug: metformin
- TLC + CZT capsules group (Experimental): transform life custom (TLC) combined with 2.52 Compound Zhenzhu Tiaozhi capsules (four tablets), PO tid
  Interventions: Dietary Supplement: TLC; Drug: Compound Zhenzhu Tiaozhi capsule
- TLC + simvastatin group (Active Comparator): transform life custom (TLC) combined with 20mg simvastatin, PO qn
  Interventions: Dietary Supplement: TLC; Drug: Simvastatin

INTERVENTIONS:
Dietary Supplement: TLC — transform life custom (TLC)
Drug: metformin — 0.5g metformin group，PO tid
  Arms: TLC + metformin group
Drug: Compound Zhenzhu Tiaozhi capsule — Compound Zhenzhu Tiaozhi capsules consist of eight Chinese herbal medications, such as Ligustrum lucidum, Atractylodes macrocephala, Radix Salviae Miltiorrhizae, pseudo-ginseng, Astragalus membranaceus.
  Arms: TLC + CZT capsules group
Drug: Simvastatin — 20mg simvastatin, PO qn
  Arms: TLC + simvastatin group

SUMMARY:
This is a randomised clinical trial which aims to evaluate the efficacy of Compound Zhenzhu Tiaozhi capsules in the treatment of NAFLD and analyze the relationship between improvement in NAFLD parameters and changes in intestinal functions.

DETAILED DESCRIPTION:
This is a randomised clinical trial which aims to evaluate the efficacy of Compound Zhenzhu Tiaozhi capsules in the treatment of NAFLD and analyze the relationship between improvement in NAFLD parameters and changes in intestinal functions. In this study, the investigators will (1)evaluate the relationship between the function of intestinal mucosal barrier, SIBO, and NAFLD;(2)assess the effects of Compound Zhenzhu Tiaozhi capsules on intrahepatic fat content, hepatic noninvasive score, liver biochemical parameters, blood lipid, and insulin resistance. To evaluate the therapeutic effects of Compound Zhenzhu Tiaozhi capsules on the treatment of NAFLD, and determine whether the risk stratification of atherosclerotic cardiovascular disease (ASCVD) and quality of life (using the 36-Item Short Form Health Survey [SF-36]) can be improved in NAFLD patients with Compound Zhenzhu Tiaozhi capsules;(3) compare the therapeutic effects of Compound Zhenzhu Tiaozhi capsules with conventional medications in the treatment of NAFLD, and to compare their efficacies in improving the risk stratification of ASCVD and quality of life, as assessed by the SF-36; (4) analyze the relationship of Compound Zhenzhu Tiaozhi capsules in improving NAFLD and parameters related to the function of the intestinal mucosal barrier and SIBO.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of simple steatosis or NASH 18 to 75 years old serum alanine transaminase (ALT)≤2 times the upper limit of normal

Exclusion Criteria:

other chronic liver diseases serious complications in other organs malignant tumors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2017-12-31 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Fat attenuation index | at 6 months following therapy
  The fat attenuation index will be used to assess the therapeutic efficacy. A normal fat attenuation index is defined as < 240 db/m, mild is 240-264 db/m, moderate is 265-294 db/m, and severity is > 295 db/m.We will detect the fat attenuation index at 6 months following treatment. Effective: fat attenuation index is reduced by a level or more (example: moderate to mild). Invalid: fails to meet the effective standard.

SECONDARY OUTCOMES:
Serum triglyceride | at 6 months following therapy
  detecting the serum level of triglyceride
Serum cholesterol | at 6 months following therapy
  detecting the serum level of cholesterol
Serum lipoproteins | at 6 months following therapy
  including chylomicron (CM), very-low-density lipoprotein (VLDL), low-density lipoprotein (LDL), and high-density lipoprotein (HDL).
Hydrogen/methane breath testing | at 6 months following therapy
  breath testing for SIBO
Quality of life | at 6 months following therapy
  The quality of life of the patients before and after treatment will be assessed using the 36-Item Short Form Health Survey and compared to assess the improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (3):
  • Study Protocol (2017-11-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03375580/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03375580/SAP_001.pdf
  • Informed Consent Form (2017-11-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03375580/ICF_002.pdf